CLINICAL TRIAL: NCT04890483
Title: Transcranial Direct Current Stimulation in Post-Acute COVID-19 Patients With Systemic Autoimmune Rheumatic Diseases
Brief Title: tDCS in Post-Acute COVID-19 Patients With SARDs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Samuel Katsuyuki Shinjo, PhD, Professor, PhD, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYO-HCFMUSP-09
Record Dates: First submitted 2021-05-17; First posted 2021-05-18 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Rheumatic Diseases; Autoimmune Diseases
MeSH Terms: conditions — Rheumatic Diseases; Autoimmune Diseases | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: An open-label uncontrolled study of application of tDCS sessions in ARD patients with post-acute COVID-19.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The ARD patients with post-acute COVID-19 will receive tDCS sessions for one week.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — tDCS: the energy of the anode (transcranial current stimulation) will have as its source a battery-powered DC generator and will be exerted by two electrodes measuring 5x7cm and attached to the head. The electrodes will be located of the primary motor cortex. The electrode with positive charge (anode) will be positioned at contralateral to the dominant limb and the negative charged electrode will be positioned in the supraorbital region ipsilateral to the dominant limb. The active current of direct transcranial stimulation will be applied with the intensity of electric current of 2mA and density of 0.057 mA/cm2 with duration of 20 minutes. During the session, patients will remain seated. Number of sessions: five times, once per day.

SUMMARY:
Some patients develop "Post-acute COVID-19 syndrome," in which they experience persistent symptoms after recovering from the acute phase of COVID-19 infection. This syndrome may be more significant in patients with systemic autoimmune rheumatic diseases (SARDs) who have been suffering from several symptoms associated to SARDs, such as myalgia, fatigue, and general pains.

The transcranial direct current stimulation (tDCS) technique has been frequent, for example, to relieve fatigue and general pains in general population. However, to date, there are no studies evaluating this technique in ARD patients with post-acute COVID-19; therefore, the main objective of the opened study is to evaluate the safety and efficacy of the application of acute tDCS in ARD patients with post-acute COVID-19.

DETAILED DESCRIPTION:
Currently, there are no studies evaluating the tDCS technique in ARD patients with post-acute COVID-19; therefore, the main objective of the present study is to evaluate the safety and efficacy of the application of acute tDCS in these specific patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with well-defined ARDs (rheumatoid arthritis, sclerosis systemic, Sjögren syndrome, spondyloarthritis, systemic lupus erythematosus, systemic vasculitis, and systemic autoimmune myopathies)
* Fatigue or general pains.

Exclusion Criteria:

* Neoplasia, using heart pacemarker, using visceral metalic clips, infections (HIV, HTLV-1, hepatitis), pregnance, previous historical of convulsions or epilepsies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-12-04 (Estimated)

PRIMARY OUTCOMES:
Frequency of treatment-emergent adverse events [safety and tolerability] | [Time Frame: After 30 minutes of transcranial stimulation.]
  Frequency of disease relapsing (based on the questionnaire of secondary outcome measures) and tolerability (patients' symptom registration)
Frequency of treatment-emergent adverse events [safety and tolerability] | [Time Frame: After 5 sessions of transcranial stimulation.]
  Frequency of disease relapsing (based on the questionnaire of secondary outcome measures) and tolerability (patients' symptom registration)
Frequency of treatment-emergent adverse events [safety and tolerability] | [Time Frame: After 30 days of transcranial stimulation.]
  Frequency of disease relapsing (based on the questionnaire of secondary outcome measures) and tolerability (patients' symptom registration)
Frequency of treatment-emergent adverse events [safety and tolerability] | [Time Frame: After 60 days of transcranial stimulation.]
  Frequency of disease relapsing (based on the questionnaire of secondary outcome measures) and tolerability (patients' symptom registration)

SECONDARY OUTCOMES:
Health Assessment Questionnaire (HAQ) | [Time Frame: 3 times: (a) within 30 minutes before stimulation. Then, after (b) one and (c) two months after stimulation]
  Especific questionnaire (health assessment questionnaire). Pontuaction 0.00 (best) - 3.00 (worst)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel K Shinjo, PhD, Principal Investigator — Sao Paulo University
Locations (1):
- Samuel K Shinjo, São Paulo, Brazil